CLINICAL TRIAL: NCT04544813
Title: A Phase 1 Study to Investigate the Pharmacokinetics and Pharmacodynamics of JNJ-77474462 in Healthy Participants
Brief Title: A Study of JNJ-77474462 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR108771; 77474462ADM1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-09-09; First posted 2020-09-10 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Healthy
MeSH Terms: interventions — bermekimab; Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Cohort A: JNJ-77474462 SC (Wave 1) (Experimental): Participants will receive single dose of JNJ-77474462 subcutaneously (SC).
  Interventions: Drug: JNJ-77474462
- Cohort B: JNJ-77474462 SC (Wave 1) (Experimental): Participants will receive single dose of JNJ-77474462 SC.
  Interventions: Drug: JNJ-77474462
- Cohort C: JNJ-77474462 SC (Wave 1) (Experimental): Participants will receive single dose of JNJ-77474462 SC.
  Interventions: Drug: JNJ-77474462
- Cohort D: JNJ-77474462 SC (Wave 1) (Experimental): Participants will receive single dose of JNJ-77474462 SC.
  Interventions: Drug: JNJ-77474462
- Cohort E: JNJ-77474462 IV (Wave 1) (Experimental): Participants will receive single dose of JNJ-77474462 intravenously (IV).
  Interventions: Drug: JNJ-77474462
- Cohort F: JNJ-77474462 SC (Wave 2) (Experimental): Participants will receive single dose of JNJ-77474462 SC.
  Interventions: Drug: JNJ-77474462
- Cohort G: JNJ-77474462 SC (Wave 2) (Experimental): Participants will receive single dose of JNJ-77474462 SC.
  Interventions: Drug: JNJ-77474462
- Cohort H: JNJ-77474462 IV (Wave 2) (Experimental): Participants will receive single dose of JNJ-77474462 IV.
  Interventions: Drug: JNJ-77474462
- Cohort I: JNJ-77474462 IV (Wave 2) (Experimental): Participants will receive single dose of JNJ-77474462 IV.
  Interventions: Drug: JNJ-77474462
- Cohort J: Anakinra SC (Active Comparator): Participants will receive a SC injection of anakinra once daily for 3 days.
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: JNJ-77474462 — Participants will receive JNJ-77474462 as a liquid formulation in Cohort A, B, C, D, F and G (SC injection) and in Cohort E, H and I (IV infusion).
  Other Names: Bermekimab
  Arms: Cohort A: JNJ-77474462 SC (Wave 1); Cohort B: JNJ-77474462 SC (Wave 1); Cohort C: JNJ-77474462 SC (Wave 1); Cohort D: JNJ-77474462 SC (Wave 1); Cohort E: JNJ-77474462 IV (Wave 1); Cohort F: JNJ-77474462 SC (Wave 2); Cohort G: JNJ-77474462 SC (Wave 2); Cohort H: JNJ-77474462 IV (Wave 2); Cohort I: JNJ-77474462 IV (Wave 2)
Drug: Anakinra — Participants will receive a SC injection of anakinra 100 mg once daily for 3 days.
  Arms: Cohort J: Anakinra SC

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (PK) of JNJ-77474462 after single subcutaneous (SC) or intravenous (IV) administrations and the effect of formulation concentrations on PK of JNJ-77474462 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy on the basis of physical examination, medical history, vital signs, and 12 lead electrocardiogram (ECG) performed at screening. Any abnormalities must be considered not clinically significant and this determination must be recorded in the participant's source documents and initialed by the investigator
* Otherwise healthy on the basis of clinical laboratory tests performed at screening and Day 1. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* A woman of childbearing potential must have a negative highly sensitive serum beta-human chorionic gonadotropin (beta hCG) at screening and a negative urine pregnancy test on Day -1
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for a period of 90 days post study intervention administration
* A male participant must agree not to donate sperm for the purpose of reproduction during the study and for a minimum of 90 days after receiving the last dose of study intervention

Exclusion Criteria:

* History of any clinically significant medical illness or medical disorders the investigator considers should exclude the participant, including (but not limited to), neuromuscular, hematological disease, immune deficiency state, respiratory disease, hepatic or gastrointestinal disease, neurological or psychiatric disease, ophthalmological disorders, neoplastic disease, renal or urinary tract diseases, or dermatological disease
* Has a history of malignancy before screening. Exceptions are squamous and basal cell carcinomas of the skin, carcinoma in situ of the cervix, or a malignancy which is considered cured with minimal risk of recurrence
* Has or has had a serious infection (example: sepsis, pneumonia, or pyelonephritis), or have been hospitalized or received intravenous (IV) antibiotics for a serious infection during the 4 months prior to the screening visit
* Is currently enrolled in an investigational study or has received an investigational intervention (including investigational vaccines or devices) 5 half-lives or 8 weeks prior to screening (whichever is longer)
* Has received prescription medications within 2 weeks prior to first study intervention administration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of JNJ-77474462 | Up to Week 12
  Cmax is the maximum observed plasma concentration.
Area Under the Plasma Concentration Versus Time Curve from Time Zero to Infinity with Extrapolation of the Terminal Phase (AUC[0-infinity]) of JNJ-77474462 | Up to Week 12
  AUC(0-infinity) is defined as area under the plasma concentration versus time curve from time zero to infinity with extrapolation of the terminal phase of JNJ-77474462.
Area Under the Plasma Concentration Versus Time Curve from Time Zero to the Time Corresponding to the Last Quantifiable Concentration (AUC[0-last]) of JNJ-77474462 | Up to Week 12
  AUC(0-last) is defined as area under the plasma concentration versus time curve from time zero to the time corresponding to the last quantifiable concentration of JNJ-77474462.
Terminal Half-Life (T1/2) of JNJ-77474462 | Up to Week 12
  T1/2 is defined as the time measured for the plasma concentration to decrease by 1 half of its original concentration.
Absolute Subcutaneous (SC) Bioavailability (F%) | Up to Week 12
  (F%) is defined as absolute SC bioavailability to be calculated using the following equation: AUC(0-infinity) SC/mean AUC(0-infinity) IV * 100 percent (%).

SECONDARY OUTCOMES:
Percentage of Participants with Treatment-emergent Adverse Events (TEAE) | Up to Week 12
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are defined as adverse events (AEs) with onset or worsening on or after date of first dose of study treatment.
Percentage of Participants with Serious Adverse Events (SAE) | Up to Week 12
  A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Number of Participants with Clinically Significant Changes in Vital Signs | Up to Week 12
  Number of participants with clinically significant changes in vital signs (including body temperature, resting [supine] pulse/heart rate, respiratory rate and blood pressure) will be reported.
Number of Participants with Clinically Significant Changes in Electrocardiogram (ECG) | Up to Week 12
  Number of participants with clinically significant changes ECG will be reported.
Number of Participants with Clinically Significant Changes in Laboratory Findings | Up to Week 12
  Number of participants with clinically significant changes in laboratory findings (that is, hematology, clinical chemistry, urinalysis) will be reported.
Number of Participants with Anti-JNJ-77474462 Antibodies | Up to Week 12
  Number of participants with anti-drug antibodies to JNJ-77474462 will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Nucleus Network, Q-Pharm Pty Ltd, Herston, Australia

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency